CLINICAL TRIAL: NCT06251856
Title: Development and Evaluation of the Effectiveness of Lower Extremity Lymphedema Education Program After Gynecological Cancer Surgery
Brief Title: Feasibility and Effectiveness of Lymphedema Education Program After Gynecological Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023.395.IRB3.172
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Lower Extremity Lymphedema
Keywords: lower limb lymphedema; gynecologic cancer surgery; quality of life; self-efficacy; symptom management model; patient education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lymphedema education (Experimental): Participants will receive lymphedema education and educational brochures from the researcher on the 2nd day after gynecological cancer surgery.
  Interventions: Behavioral: lymphedema education program
- routine discharge education (No Intervention): Routine post-op discharge education is given to patients who undergo gynecological cancer surgery at the institution by nurses on the day of discharge.

INTERVENTIONS:
Behavioral: lymphedema education program — On post-op day 2, patients will receive Symptom Management Model-Based Lower Extremity Lymphedema Training. Brochures will be introduced and delivered to the patient.
  Arms: lymphedema education

SUMMARY:
This study aims to examine the effect of lower extremity lymphedema prevention training based on the Symptom Management Model on women undergoing gynecological cancer surgery on lymphedema development, quality of life, and women's self-efficacy. The hypotheses of the study are:

H1a: The quality of life of women who underwent gynecological cancer surgery and received lower extremity lymphedema prevention training based on the Symptom Management Model is statistically significantly higher than the quality of life of women in the control group.

H1b: The self-efficacy levels of women who underwent gynecological cancer surgery and received lower extremity lymphedema prevention training based on the Symptom Management Model are statistically significantly higher than the self-efficacy levels of women in the control group.

H1c: The frequency of experiencing lower extremity lymphedema symptoms of women who underwent gynecological cancer surgery and received lower extremity lymphedema prevention training based on the Symptom Management Model is significantly lower than the frequency of experiencing lower extremity lymphedema symptoms of women in the control group.

Participants will be given training on lower extremity lymphedema. At the end of the study, researchers will evaluate the impact of the training on quality of life, self-efficacy, and lymphedema development.

DETAILED DESCRIPTION:
The incidence of lower extremity lymphedema following gynecological cancer treatment varies depending on the type of gynecological cancer. The prevalence of lymphedema varies between 1-38% in endometrial cancers, 17-81% in cervical cancers, 6-75% in vulvar-vaginal cancers, and 5-21% in ovarian cancers. Studies have shown that the risk of developing lymphedema after gynecological cancer persists in the long term, although the majority of cases occur in the first year. The main factors that increase the risk of developing lower extremity lymphedema are stated as Body Mass Index (BMI), age, The International Federation of Gynecology and Obstetrics (FIGO) cancer stage, lymph node dissection and number of lymph nodes. Lower extremity lymphedema is characterized by symptoms such as unilateral or bilateral swelling, heaviness, pain, itching, numbness, skin changes, infection, etc. These symptoms can seriously affect the patient's quality of life by limiting their daily living activities. Therefore, there is a need for effective interventions to prevent and manage lower extremity lymphedema associated with cancer treatment to improve quality of life and well-being. The training is planned to be structured according to the Symptom Management Model. After gynecological cancer surgery, women's ability to self-diagnose the symptoms they experience related to lymphedema and their responses to these symptoms become part of the management process. In this regard, it is thought that nurse-led education programs positioned in a theoretical framework to prevent lower extremity lymphedema will enable patients to diagnose the early symptoms of lymphedema by improving their knowledge, quality of life, self-efficacy, and reduce the risk of lymphedema. It is anticipated that the model-based nurse-led education program to be developed in this study will be applicable in the clinic and the evidence obtained will guide future research. After obtaining institutional permission, data will be collected by the researcher through a face-to-face interview with women over the age of 18 who meet the inclusion criteria. During this visit, face-to-face information about the research will be given, written consent will be obtained, and data collection tools will be introduced and filled in. The risks of the participants will be determined with the lymphedema risk assessment questionnaire and stratified randomization will be provided accordingly. Research data will be collected with the Socio-demographic Information Form, the Information Form on Cancer Diagnosis, the Lymphedema Risk Assessment Questionnaire, the European Organization for Research and Treatment of Cancer Quality of Life Scale, the 6-Item Self-Efficacy Scale for Chronic Disease Management, Gynecological Cancer Lymphedema Questionnaire and Lower extremity circumference measurement. After data collection, the data will be transferred to the Statistical Package for the Social Sciences (SPSS) 26.0 software package for analysis. The data analysis will include percentages, mean values, standard deviations and chi-square test, independent sample t-test, repeated measures ANOVA test, and the corrected Bonferroni test for advanced analyses.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age,
* Able to speak and understand Turkish,
* Not having any cognitive, visual or auditory disabilities,
* Diagnosed with gynecological cancer (cervix, ovary, uterus, endometrium, vulva, etc.)
* Women who underwent gynecological surgery with inguinal and/or para-aortic and/or pelvic lymph node dissection due to malignancy.
* Women who have accepted and signed the consent and consent document

Exclusion Criteria:

* Women who diagnosed with venous insufficiency and peripheral artery disease,
* Women with previously diagnosed lower extremity lymphedema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Gynecological Cancer Lymphedema Questionnaire (GCLQ)- experiences of lymphedema symptoms | 3th month and 6th month
  The scale questions are answered with a "yes" or "no". GCLQ contains 20 questions that evaluate the presence of symptoms over the past four weeks, scored as 0. If a patient scores 20 points on GCLQ, it indicates the presence of all symptoms, while a score of 0 indicates the absence of all symptoms.
Lower Extremity Circumference Measurement | baseline, 3th and 6th month
  Circumference measurements will be taken in the supine position, moving from the medial malleolus to the inguinal region at 5 cm intervals for both lower extremities. The difference between both extremities will be recorded in cm. A difference of 2 cm between sides measured from at least 6 points is considered significant.
The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) (C30-VERSION 3.0) | baseline, 3th and 6th month
  The answers are rated from "not at all" (1 point) to "a lot" (4 points). The last two questions (29th and 30th) are related to the general quality of life and ask the patient to evaluate their health and quality of life in the last week on a scale of 1 to 7 (1 being "very bad" and 7 being "very good"). High scores from these questions indicate high quality of life, while low scores indicate low quality of life.; very bad, 7 points; very good).
6-Item Self-Efficacy Scale for Chronic Disease Management | baseline, 3th and 6th month
  The scale consists of six items, with the first four measuring behavioral attitude and the last two measuring psychological attitude. Each item is rated on a 10-point scale ranging from "not at all confident" to "completely confident." To obtain the score, the average of all six items is calculated, with higher scores indicating greater self-efficacy.

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Abakay H, Abdulrezzak U, Akbayrak T. (2022). An Important Tool in Lymphedema Management: Validation of the Turkish Version of the Gynecologic Cancer Lymphedema Questionnaire. Gynecol Obstet Reprod Med. https://doi.org/10.21613/GORM.2022.1348
- [Background] Backler C, Beck M, Poage E. Lymphedema: Clinical Summary of the ONS Guidelines for Cancer Treatment-Related Lymphedema. Clin J Oncol Nurs. 2020 Oct 1;24(5):566-570. doi: 10.1188/20.CJON.566-570. PMID 32945785
- [Background] Bakar Y, Tugral A. Lower Extremity Lymphedema Management after Gynecologic Cancer Surgery: A Review of Current Management Strategies. Ann Vasc Surg. 2017 Oct;44:442-450. doi: 10.1016/j.avsg.2017.03.197. Epub 2017 May 5. PMID 28483624
- [Background] Hayes SC, Janda M, Ward LC, Reul-Hirche H, Steele ML, Carter J, Quinn M, Cornish B, Obermair A. Lymphedema following gynecological cancer: Results from a prospective, longitudinal cohort study on prevalence, incidence and risk factors. Gynecol Oncol. 2017 Sep;146(3):623-629. doi: 10.1016/j.ygyno.2017.06.004. Epub 2017 Jun 16. PMID 28624154
- [Background] Bowman C, Piedalue KA, Baydoun M, Carlson LE. The Quality of Life and Psychosocial Implications of Cancer-Related Lower-Extremity Lymphedema: A Systematic Review of the Literature. J Clin Med. 2020 Oct 2;9(10):3200. doi: 10.3390/jcm9103200. PMID 33023211
- [Background] Cal A, Bahar Z, Gorken I. Effects of Health Belief Model based nursing interventions offered at home visits on lymphedema prevention in women with breast cancer: A randomised controlled trial. J Clin Nurs. 2020 Jul;29(13-14):2521-2534. doi: 10.1111/jocn.15271. Epub 2020 Apr 17. PMID 32243029
- [Background] Cankurtaran ES, Ozalp E, Soygur H, Ozer S, Akbiyik DI, Bottomley A. Understanding the reliability and validity of the EORTC QLQ-C30 in Turkish cancer patients. Eur J Cancer Care (Engl). 2008 Jan;17(1):98-104. doi: 10.1111/j.1365-2354.2007.00827.x. PMID 18181898
- [Background] Deura I, Shimada M, Hirashita K, Sugimura M, Sato S, Sato S, Oishi T, Itamochi H, Harada T, Kigawa J. Incidence and risk factors for lower limb lymphedema after gynecologic cancer surgery with initiation of periodic complex decongestive physiotherapy. Int J Clin Oncol. 2015 Jun;20(3):556-60. doi: 10.1007/s10147-014-0724-0. Epub 2014 Jul 4. PMID 24993674
- [Background] Do JH, Choi KH, Ahn JS, Jeon JY. Effects of a complex rehabilitation program on edema status, physical function, and quality of life in lower-limb lymphedema after gynecological cancer surgery. Gynecol Oncol. 2017 Nov;147(2):450-455. doi: 10.1016/j.ygyno.2017.09.003. Epub 2017 Sep 20. PMID 28941657
- [Background] Incirkus K, Nahcivan N. Validity and reliability study of the Turkish version of the self-efficacy for managing chronic disease 6-item scale. Turk J Med Sci. 2020 Aug 26;50(5):1254-1261. doi: 10.3906/sag-1910-13. PMID 32336077